CLINICAL TRIAL: NCT03855566
Title: Telenutrition Center: Examining the Implementation of Behavioral Therapy for Obesity Among Young to Middle Aged African American Adults in Mississippi
Brief Title: Telenutrition Center: Examining the Implementation of Behavioral Therapy for Obesity
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The study was disrupted by and results confounded by the COVID-19 pandemic and there it was not possible to meet study goals within the required timeframe.
Sponsor: University of Southern Mississippi (Other)
Collaborators: My Brother's Keeper, Inc. (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P20GM103476 (NIH)
Record Dates: First submitted 2019-02-21; First posted 2019-02-26 (Actual); Last update posted 2023-07-18 (Actual); Status verified 2023-07

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — Adiposity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Other): Enrolled participants will receive the intervention.
  Interventions: Behavioral: Intensive behavioral therapy for obesity

INTERVENTIONS:
Behavioral: Intensive behavioral therapy for obesity — Approximately 24, 20 minute sessions over 12 months focused on diet and physical activity behavior change goals to promote weight loss. Framework includes health belief model, transtheoretical model and motivational interviewing.

SUMMARY:
The Telenutrition Center will use the Reach, Effectiveness, Adoption, Implementation and Maintenance (RE-AIM) Framework to assess the implementation of an evidence-based, intensive behavior therapy (IBT) for obesity intervention (with a motivational interviewing [MI] framework) based on the Centers for Medicaid and Medicare Services (CMS) IBT for obesity benefit. The intervention will be examined under real-world conditions with technology supplementation to address obesity and related chronic disease among young adult (18-50 years of age) African Americans across the state. The intervention contact will model the CMS IBT for obesity benefit according to the patient contact schedule (of weekly visits in the first month, biweekly in months 2-7, and once a month per months 8-12) and include nutrition, stage of change and other physical and psychosocial assessments. Program delivery will be assisted by the "Bridge2U" web and mobile platform and supported in both clinic and community settings. The proposed project will shed new light on how IBT for obesity (and similar) models may be amended to facilitate the provision of health care resources in areas with limited to no resources, such as the state of Mississippi.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index >/=28
* 25 to 50 years of age
* history or risk of preventable co-morbidities (ie. diabetes, hypertension, and/or dyslipidemia)

Exclusion Criteria:

* Body mass index <28
* <25 years of age
* >50 years of age
* no history or risk of preventable obesity comorbidities
* Any disease diagnosis (ie. cancer) where weight loss is contraindicated

Ages: 25 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2023-05-31 (Actual); Study Completion 2023-05-31 (Actual)

PRIMARY OUTCOMES:
Weight Changes | 0, 6 and 12 months
  Weight loss at 0, 6 and 12 months
Retention | 12 months
  Number of enrolled participants who complete the program

CONTACTS AND LOCATIONS:
Locations (1):
- The University of Southern Mississippi, Hattiesburg, Mississippi, United States